CLINICAL TRIAL: NCT01276665
Title: Effects of Noradrenaline Administration Combined With Restrictive Intraoperative Fluid Substitution on Blood Loss and Perioperative Outcome in Patients Undergoing Open Radical Cystectomy
Brief Title: Effects of Noradrenaline Administration Combined With Restrictive Intraoperative Fluid Substitution on Perioperative Outcome in Patients Undergoing Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Dr Patrick Wüthrich/Department of Anesthesiology and Pain Therapy, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 154/08
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Bladder Cancer; Urinary Diversion
Keywords: Bladder cancer; urinary diversion; Postoperative Complications; Fluid Therapy; Norepinephrine
MeSH Terms: conditions — Urinary Bladder Neoplasms; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restrictive regimen group (Experimental): treated with a restrictive fluid regimen of 2ml/kg/h of crystalloids in combination with sympathicomimetics.
  Interventions: Procedure: restrictive intraoperative fluid substitution
- Control group (Active Comparator): treated according to an internationally accepted standard fluid regimen (6 ml/kg/h of crystalloids and correction of the hypotony with fluid boluses)
  Interventions: Procedure: assessment of the pelvic venous pressure

INTERVENTIONS:
Procedure: restrictive intraoperative fluid substitution — to analyze the impact of a restrictive volume regimen using advanced balanced electrolyte solution (which is by far more restrictive than the published data) combined with noradrenaline. We include only radical cystectomy and so nearly exclude surgical bias
  Arms: Restrictive regimen group
Procedure: assessment of the pelvic venous pressure — A 20 G catheter will be introduced into a small collateral vein of the internal iliacal vein to monitor pelvic venous pressure
  Arms: Control group

SUMMARY:
Perioperative fluid management in abdominal surgery is a subject of controversy and current standard fluid therapy is not evidence based. Compensating decreasing blood pressure by volume substitution is common praxis. Alternatively the fall in blood pressure due to vasodilatation can be corrected by applying vasoactive agents. A review of the data on the effect of "high volume" perioperative fluid therapy suggests that overhydration may have deleterious effects on cardiopulmonary function as well as on recovery of gastrointestinal motility, tissue oxygenation and wound healing. Restrictive fluid administration in fast-track surgery led to no differences in all-over recovery after colonic surgery. Based on our current knowledge, a low volume regimen combined with a noradrenaline perfusor may be of benefit during open radical cystectomy. It seems of interest and safe to use a noradrenaline perfusor combined with a low volume regimen during open radical cystectomy. The low volume regimen, as described in this study protocol, is well established at our institution, which has a large experience in cystectomy.

The aim of this study is to compare intraoperative blood loss, quality of the surgical field, metabolic response, pain relief, fatigue score, gastrointestinal function, cardiovascular, pulmonary, infectious and surgical complications as well as cognitive function in two groups of patients undergoing radical cystectomy.

The investigators expect a lower complication rate in the restrictive fluid regimen group and better surgical conditions. This could significantly affect short- and long-term outcome of patient undergoing major cancer surgery, have an impact on survival and financial consequences.

DETAILED DESCRIPTION:
Background

Perioperative fluid management in abdominal surgery is a subject of controversy and current standard fluid therapy is not evidence based. Standard fluid therapy includes replacement of basic fluid requirements, loss by perspiration, by exsudation through the surgical wound, and loss into the third space.

Fluid preload before spinal or just after epidural anaesthesia is a common and recognized practice in clinical anaesthesia. Vasodilatation is a well-known side effect of halogenics, of most hypnotics and opiates. Compensating decreasing blood pressure by volume substitution is common praxis. Alternatively the fall in blood pressure due to vasodilatation can be corrected by applying vasoactive agents. A review of the data on the effect of "high volume" perioperative fluid therapy suggests that overhydration may have deleterious effects on cardiopulmonary function (excessive shift to the right on the Starling myocardial performance curve, pneumonia and respiratory failure) as well as on recovery of gastrointestinal motility (prolonged postoperative ileus (PI)), tissue oxygenation and wound healing (anastomosis leakage). A postoperative weight gain of 3-7 kg in patients after major elective surgery therefore seems to represent a genuine fluid overload. Delay in bowel motility may be due to the presence of excess fluid in the intestinal wall resulting from excess perioperative fluid therapy. Increased gut permeability after surgical trauma may also contribute to the development of PI because of enhanced uptake of luminal bacterial products. Postoperative complications were significantly reduced by restricted fluid therapy. A dose response relation between administrated fluid volume and postoperative complications (cardiopulmonary and tissue healing) was found in a randomised assessor blinded multicenter trial for colorectal surgery 11,12. The restricted fluid regimen did not lead to haemodynamic instability and the amount of vasoactive substances administered was similar. No significant difference in urinary output was demonstrated on days 1 and 6. Restrictive fluid administration in fast-track surgery led to no differences in all-over recovery after colonic surgery. Goal-directed intraoperative fluid administration using the oesophageal Doppler monitor to maintain maximal stroke volume has been shown to reduce the length of hospital stay, lower the incidence of postoperative nausea and vomiting and to encourage an early return of bowel function. Oesophageal Doppler monitor permits rapid, minimally invasive and continuous estimation of cardiac output. It can be easily inserted and is not associated with major complications. The investigators will use oesophageal Doppler monitoring for intraoperative monitoring of stroke volume and cardiac output.

In animal experiments on pigs, high (18ml/kg/h) or low (3ml/kg/h) volume crystalloid fluid treatment had no effect on colon tissue oxygenation tension. Three different fluid volume regimens (3ml/kg/h, 7 ml/kg/h and 20ml/kg/h) tested did not affect tissue oxygen pressure in the jejunum and colon, suggesting efficient autoregulation of intestinal blood flow in healthy pigs undergoing uncomplicated abdominal surgery 25. Noradrenaline increased systemic blood flow (mean arterial pressure and cardiac index) and failed to increase microcirculatory blood flow in most abdominal organs in septic pigs. Thoracic epidural anesthesia per se does not affect intravascular volume. Therefore, vasopressors are preferable for treatment of hypotension after epidural anesthesia.

The incidence of postoperative cognitive dysfunction varies greatly with reported rates of 10% to 55%. Patient characteristics such as age, education, type and length of surgical procedure and preoperative cognitive status have been found to affect the incidence and severity of postoperative cognitive dysfunction. The influence of intraoperative volume management on cognitive function has not been assessed.

It seems of interest and safe to use a noradrenaline perfusor combined with a low volume regimen during open radical cystectomy. The low volume regimen, as described in this study protocol, is well established in our institution, which has a large experience in cystectomy.

Objective

The aim of this study is to compare intraoperative blood loss, quality of the surgical field (defined later), metabolic response, pain relief, fatigue score, gastrointestinal function, cardiovascular, pulmonary, infectious and surgical complications and cognitive function in two groups of patients undergoing radical cystectomy. The first group will be treated according to an internationally accepted standard fluid regimen (6 ml/kg/h of crystalloids and correction of the hypotony with fluid boluses); the second one will be treated with a restrictive fluid regimen of 2ml/kg/h of crystalloids in combination with sympathicomimetics.

Methods

Prospective, randomised, controlled, single-centre study. Randomly assigned in equal proportion by computer to receive the dry regimen 2ml/kg/h combined with sympathicomimetics or the standard fluid management.

An advanced balanced electrolyte solution will be used containing acetate/malate instead of lactate. Substantial advantages are a base excess of +/- O mmol/l, that it is isotonic, and contains anions acetate and malate.

208 patients with open radical cystectomy Duration: 36 months Setting: University Department of Urology , Inselspital Bern, Switzerland Study sample and power calculation

A power analysis for postoperative complication rate as primary outcome has been done with the NCSS PASS programme:

Power: 80% Significance: 0.05% or lower Complication rate for the restrictive volume regimen group: 20% Complication rate for the control group: 38% 83 patients will be required in each group. Assuming a 20% drop-out rate 104 patients per group will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* ASA 1 to 3
* Radical cystectomy with ileal neobladder/ileum conduit

Exclusion Criteria

* Coagulopathies
* - Significant hepatic dysfunction (liver enzymes > 50% upper normal value)
* - Significant renal dysfunction: GFR< 60 ml/min/1,73 m² (Kidney Disease Outcomes Quality Initiative stade 3 or more )
* Congestive heart failure
* Oesophageal pathology
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Complications (morbidity score) | during hospitalisation, at 30 days postoperative

SECONDARY OUTCOMES:
Perioperative blood loss and quality of the surgical field | intraoperative
-Hospital stay | hospital discharge
Correlation between pelvic venous pressure and bleeding | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wuethrich, MD, Principal Investigator — Dep. of Anesthesiology and Pain Therapy, University Hospital Beern, Switzerland
Locations (1):
- Dep. of Anesthesiology and Pain Therapy, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Nisanevich V, Felsenstein I, Almogy G, Weissman C, Einav S, Matot I. Effect of intraoperative fluid management on outcome after intraabdominal surgery. Anesthesiology. 2005 Jul;103(1):25-32. doi: 10.1097/00000542-200507000-00008. PMID 15983453